CLINICAL TRIAL: NCT03155386
Title: Evaluation of the Clinical Performance of Optimized Angiomammography and Comparison With Standard Angiomammography
Brief Title: Optimized Angiomammography and Comparison With Standard Angiomammography
Acronym: OPTIAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-A01566-45; 2016/2643 (Other: CSET number)
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Patients for Whom an Angiomammogram Examination is Requested Whether Its Indication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard Angiomammography (SenoBright®)
  Interventions: Other: Angiommamography
- Optimized angiomammography
  Interventions: Other: Angiommamography

INTERVENTIONS:
Other: Angiommamography — A blinded central re-reading of the acquisition technique will be carried out by 3 radiologists (2 seniors and 1 junior) who will evaluate:
  * The intensity of lesion enhancement
  * The presence and type of artefacts on the recombined images.
  * The quality of low-energy images according to recognized criteria for mammography.
  The gold standard will be histology (biopsies or surgery) or follow-up to 1 year for non-biopsied benign lesions

SUMMARY:
This study will be proposed consecutively to any patient who angiomammography examination was requested by the clinician in charge of patient. A randomization will be performed between an angiomammography examination Standard (SenoBright®) and an optimized angiomammography examination.

A blinded central re-reading of the acquisition technique will be carried out by 3 radiologists (2 seniors and 1 junior) who will evaluate:

* The intensity of lesion enhancement
* The presence and type of artefacts on the recombined images.
* The quality of low-energy images according to recognized criteria for mammography.

The gold standard will be histology (biopsies or surgery) or follow-up to 1 year for non-biopsied benign lesions

ELIGIBILITY:
Inclusion Criteria:

1. Patient for whom angiomammography examination is requested regardless of its indication (assessment of extension, clarification of a lesion doubtful after mammography and mammary ultrasound, symptom mammary MRI in a patient with contraindication to MRI)
2. Patient aged 40 to 70 years
3. Informing the patient or his / her legal representative and signing the form of non-opposition.
4. Patient affiliated to a social security system.

Exclusion Criteria:

1. Patient with breast prostheses
2. Patient with a genetic mutation (BRCA1, BRCA2, p57)
3. Contraindication to injection of iodinated contrast agent
4. Pregnant woman, likely to be pregnant or breastfeeding,
5. Persons deprived of their liberty or under guardianship,
6. Unable to undergo medical follow-up of the trial for reasons geographical, social or psychological.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients for whom an angiomammographic examination is requested regardless of its indication
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05-18 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
artefact presence rate | up to 12 months
  Compare the artefact presence rate per patient for optimized angiomammography images and images of the Senobright® product.

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val de Marne, France

IPD SHARING:
Plan to Share IPD: Undecided